CLINICAL TRIAL: NCT03298451
Title: A Randomized, Open-label, Multi-center Phase III Study of Durvalumab and Tremelimumab as First-line Treatment in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Study of Durvalumab and Tremelimumab as First-line Treatment in Patients With Advanced Hepatocellular Carcinoma
Acronym: HIMALAYA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419CC00002; 2024-512212-21-00 (Registry Identifier: CTIS (EU)); 2016-005126-11 (EudraCT Number)
Record Dates: First submitted 2017-09-19; First posted 2017-10-02 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma Non-Resectable
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; tremelimumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Durvalumab
  Interventions: Drug: Durvalumab
- Arm 2 (Experimental): Durvalumab in combination with tremelimumab (Regimen 1)
  Interventions: Drug: Tremelimumab (Regimen 1); Drug: Durvalumab (Regimen 1)
- Arm 3 (Experimental): Durvalumab in combination with tremelimumab (Regimen 2)
  Interventions: Drug: Tremelimumab (Regimen 2); Drug: Durvalumab (Regimen 2)
- Arm 4 (Active Comparator): Sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous infusion).
  Other Names: MEDI4736
  Arms: Arm 1
Drug: Tremelimumab (Regimen 1) — Tremelimumab IV (intravenous infusion).
  Arms: Arm 2
Drug: Tremelimumab (Regimen 2) — Tremelimumab IV (intravenous infusion).
  Arms: Arm 3
Drug: Sorafenib — Sorafenib, as per standard of care
  Arms: Arm 4
Drug: Durvalumab (Regimen 1) — Durvalumab IV (intravenous infusion).
  Arms: Arm 2
Drug: Durvalumab (Regimen 2) — Durvalumab IV (intravenous infusion).
  Arms: Arm 3

SUMMARY:
This is a randomized, open-label, multi-center, global, Phase III study to assess the efficacy and safety of durvalumab plus tremelimumab combination therapy and durvalumab monotherapy versus sorafenib in the treatment of patients with no prior systemic therapy for unresectable HCC. The patients cannot be eligible for locoregional therapy

DETAILED DESCRIPTION:
The study population includes patients 18 years of age or older with advanced HCC, Barcelona Clinic Liver Cancer stage B not eligible for locoregional therapy or stage C, and Child-Pugh A classification liver disease. Patients must not have received any prior systemic therapy for unresectable HCC.

Patients in all treatment arms may continue receiving their originally assigned treatment, at the Investigator's discretion, until progression

Patients in all arms with confirmed PD who, in the Investigator's opinion, continue to receive benefit from their assigned treatment and meet the criteria for treatment in the setting of PD may continue to receive their assigned treatment.

If a patient discontinues study drug(s) due to disease progression, the patient will enter survival follow-up. Patients who have discontinued treatment due to toxicity or symptomatic deterioration or who have commenced subsequent anticancer therapy, will have tumor assessments until confirmed PD and will be followed for survival

ELIGIBILITY:
Inclusion criteria

* HCC based on histopathological confirmation
* No prior systemic therapy for HCC
* Barcelona Clinic Liver Cancer (BCLC) stage B (that is not eligible for locoregional therapy) or stage C
* Child-Pugh Score class A
* ECOG performance status of 0 or 1 at enrollment

Exclusion criteria

* Hepatic encephalopathy within past 12 months or requirement for medication to prevent or control encephalopathy
* Clinically meaningful ascites
* Main portal vein tumor thrombosis
* Active or prior documented GI bleeding (eg, esophageal varices or ulcer bleeding) within 12 months
* HBV and HVC co-infection, or HBV and Hep D co-infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1324 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2026-08-27 (Estimated)

CONTACTS AND LOCATIONS:
Locations (154):
- United States (17):
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Westwood, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Murray, Utah
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (9):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- China (18):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Dalian
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- France (14):
  - Research Site, Clichy
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Saint-Etienne
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (10):
  - Research Site, Aachen
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Tübingen
  - Research Site, Ulm
- Research Site, Hong Kong, Hong Kong
- India (9):
  - Research Site, Bangalore
  - Research Site, Bhubneshwar
  - Research Site, Chennai
  - Research Site, Hubli
  - Research Site, Hyderabad
  - Research Site, Karmsad
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, New Delhi
- Italy (8):
  - Research Site, Benevento
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (23):
  - Research Site, Bunkyoku
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Iizuka
  - Research Site, Kanazawa
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kurume
  - Research Site, Matsuyama
  - Research Site, Mitakashi
  - Research Site, Musashino
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ōgaki
  - Research Site, Ōsaka-sayama
  - Research Site, Saga
  - Research Site, Sapporo
  - Research Site, Shiwa
  - Research Site, Suntogun
  - Research Site, Tsu
  - Research Site, Yokohama
- Russia (8):
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Ufa
- South Korea (5):
  - Research Site, Ilsan, Gyeonggi-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seoul
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Pamplona Madrid
  - Research Site, Santander
- Taiwan (6):
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chang Mai
  - Research Site, Khon Kaen
  - Research Site, Phitsanulok
  - Research Site, Songkhla
- Ukraine (8):
  - Research Site, Dnipro
  - Research Site, IvanoFrankivsk
  - Research Site, Kharkiv
  - Research Site, Kropyvnitskyi
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Uzhhorod
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Hochiminh

REFERENCES:
- [Derived] Chan SL, Kudo M, Sangro B, Kelley RK, Kim JH, Pham B, Hong JY, Waldschmidt DT, Marino D, Joycelyn Lee JX, Gerolami R, Burgoyne AM, Li Q, Nakamura H, Sun P, Baur B, Rimassa L. Early Safety Results from the Phase 3b SIERRA Study of Durvalumab and Tremelimumab as First-Line Treatment for Participants with Unresectable Hepatocellular Carcinoma and a Poor Prognosis. Liver Cancer. 2025 Dec 18. doi: 10.1159/000549955. Online ahead of print. PMID 41585428
- [Derived] Rimassa L, Chan SL, Sangro B, Lau G, Kudo M, Reig M, Breder V, Ryu MH, Ostapenko Y, Sukeepaisarnjaroen W, Varela M, Tougeron D, Crysler OV, Bouattour M, Van Dao T, Tam VC, Faccio A, Furuse J, Jeng LB, Kang YK, Kelley RK, Paskow MJ, Ran D, Xynos I, Kurland JF, Negro A, Abou-Alfa GK. Five-year overall survival update from the HIMALAYA study of tremelimumab plus durvalumab in unresectable HCC. J Hepatol. 2025 Oct;83(4):899-908. doi: 10.1016/j.jhep.2025.03.033. Epub 2025 Apr 11. PMID 40222621
- [Derived] Lau G, Abou-Alfa GK, Cheng AL, Sukeepaisarnjaroen W, Van Dao T, Kang YK, Thungappa SC, Kudo M, Sangro B, Kelley RK, Furuse J, Park JW, Sunpaweravong P, Fasolo A, Yau T, Kawaoka T, Azevedo S, Reig M, Assenat E, Yarchoan M, He AR, Makowsky M, Gupta C, Negro A, Chan SL. Outcomes in the Asian subgroup of the phase III randomised HIMALAYA study of tremelimumab plus durvalumab in unresectable hepatocellular carcinoma. J Hepatol. 2025 Feb;82(2):258-267. doi: 10.1016/j.jhep.2024.07.017. Epub 2024 Jul 31. PMID 39089633
- [Derived] Sangro B, Galle PR, Kelley RK, Charoentum C, De Toni EN, Ostapenko Y, Heo J, Cheng AL, Wilson Woods A, Gupta C, Abraham J, McCoy CL, Patel N, Negro A, Vogel A, Abou-Alfa GK. Patient-Reported Outcomes From the Phase III HIMALAYA Study of Tremelimumab Plus Durvalumab in Unresectable Hepatocellular Carcinoma. J Clin Oncol. 2024 Aug 10;42(23):2790-2799. doi: 10.1200/JCO.23.01462. Epub 2024 May 28. PMID 38805668
- [Derived] Abou-Alfa GK, Lau G, Kudo M, Chan SL, Kelley RK, Furuse J, Sukeepaisarnjaroen W, Kang YK, Van Dao T, De Toni EN, Rimassa L, Breder V, Vasilyev A, Heurgue A, Tam VC, Mody K, Thungappa SC, Ostapenko Y, Yau T, Azevedo S, Varela M, Cheng AL, Qin S, Galle PR, Ali S, Marcovitz M, Makowsky M, He P, Kurland JF, Negro A, Sangro B. Tremelimumab plus Durvalumab in Unresectable Hepatocellular Carcinoma. NEJM Evid. 2022 Aug;1(8):EVIDoa2100070. doi: 10.1056/EVIDoa2100070. Epub 2022 Jun 6. PMID 38319892
- [Derived] Addendum 1: Society for Immunotherapy of Cancer (SITC) clinical practice guideline on immunotherapy for the treatment of hepatocellular carcinoma. J Immunother Cancer. 2023 Sep;11(9):e002794add1. doi: 10.1136/jitc-2021-002794add1. No abstract available. PMID 37678916
- [Derived] Patel TH, Brewer JR, Fan J, Cheng J, Shen YL, Xiang Y, Zhao H, Lemery SJ, Pazdur R, Kluetz PG, Fashoyin-Aje LA. FDA Approval Summary: Tremelimumab in Combination with Durvalumab for the Treatment of Patients with Unresectable Hepatocellular Carcinoma. Clin Cancer Res. 2024 Jan 17;30(2):269-273. doi: 10.1158/1078-0432.CCR-23-2124. PMID 37676259
- See also: CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419CC00002&attachmentIdentifier=5492a658-0cae-4a53-9c5f-2c7d7dd2f180&fileName=419CC00002CSP_redacted.pdf&versionIdentifier=
- See also: SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419CC00002&attachmentIdentifier=dfa10daf-41b0-454d-ab99-f62959a00fdc&fileName=D419CC00002_SAP_redacted.pdf&versionIdentifier=
- See also: CSR_synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419CC00002&attachmentIdentifier=7f90991f-10dd-4176-8b36-c5535f3ba6d6&fileName=D419CC00002_CSR__synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study includes 1324 participants. Participants were screened in 16 countries from Oct2017 to Jun2019. Recruitment in T75+D arm was closed during the study. Results are reported at data cut-off (DCO).
Pre-assignment Details: Of 1,950 participants screened in the study, 1,324 were randomized across 4 arms, out of which 1,302 participants received treatment.
Groups:
- Durva 1500 mg: Durvalumab 1500 mg every 4 weeks (Q4W)
- Treme 300 mg x1 Dose + Durva 1500 mg: Tremelimumab 300 mg × 1 dose + durvalumab 1500 mg Q4W
- Treme 75 mg x4 Doses + Durva 1500 mg: Tremelimumab 75 mg Q4W × 4 doses + durvalumab 1500 mg Q4W
- Sora 400 mg: Sorafenib 400 mg twice daily (BID)
Period: Overall Study
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Started (Randomized) | 389 | 393 | 153 | 389
Received Treatment (One participant in T300+D and one in T75+D arm didn't receive Treme and were analyzed under the Durva mono arm in the safety analysis set) | 386 | 389 | 153 | 374
Completed (Completed final analysis and ongoing in long-term follow-up) | 104 | 125 | 30 | 82
Not Completed | 285 | 268 | 123 | 307
Not completed — Death | 275 | 260 | 122 | 280
Not completed — Lost to Follow-up | 1 | 1 | 0 | 7
Not completed — Withdrawal by Subject | 9 | 7 | 1 | 20

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg | Total
Number analyzed (Participants) | 389 | 393 | 153 | 389 | 1324
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (11.47) | 63.0 (11.65) | 63.4 (12.03) | 63.5 (11.12) | 63.1 (11.48)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 203 | 195 | 74 | 195 | 667
  >=65-<75 | 130 | 145 | 55 | 137 | 467
  >=75 | 56 | 53 | 24 | 57 | 190
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 66 | 32 | 52 | 216
  Male | 323 | 327 | 121 | 337 | 1108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 160 | 182 | 70 | 179 | 591
  Black or African American | 2 | 7 | 4 | 10 | 23
  Asian | 212 | 195 | 75 | 189 | 671
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Other | 15 | 7 | 4 | 5 | 31
  Missing | 0 | 1 | 0 | 6 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 21 | 11 | 21 | 66
  Not Hispanic or Latino | 376 | 372 | 142 | 362 | 1252
  Missing | 0 | 0 | 0 | 6 | 6
Region group [Count of Participants; unit: Participants]
  Asia (except Japan) | 167 | 156 | 60 | 156 | 539
  Rest of World (includes Japan) | 222 | 237 | 93 | 233 | 785

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) - Treme 300 mg x1 Dose + Durva 1500 mg vs Sora 400 mg
Description: OS was defined as the time from the date of randomization until death due to any cause, regardless of whether the participant withdrew from randomized therapy or received another anticancer therapy. Any participant not known to have died at the DCO date was censored based on the last recorded date on which the participant was known to be alive. If the last known date alive or if the date of death was after the DCO date, participants were censored at the DCO date. This primary outcome measure presents OS analysis of Treme 300mg x1 dose + Durva 1500 mg vs Sora 400 mg at the time of the final analysis DCO (27Aug2021).
Time Frame: From the date of randomization until death due to any cause, assessed up to the data cut-off date (27Aug2021, to a maximum of approximately 46 months).
Population: The FAS included all participants who were randomized. T75+D arm was closed during study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 389 | 393 | 153 | 389
months | 16.56 [14.06 to 19.12] | 16.43 [14.16 to 19.58] | 16.36 [12.39 to 19.65] | 13.77 [12.25 to 16.13]
Statistical Analysis 1: Comparison: Treme 300 mg x1 Dose + Durva 1500 mg vs Sora 400 mg; The analysis was performed using stratified log-rank test adjusting for treatment, etiology of liver disease (HBV versus HCV versus others), ECOG (0 versus 1), and macro-vascular invasion (yes versus no). The values of the stratification factors were obtained from IVRS; Test type: Superiority; p = 0.0035, Log Rank — The adjusted alpha levels (0.0398) for the two-sided superiority test were derived based upon the exact number of OS events for each comparison using the Lan and DeMets approach that approximates the O'Brien Fleming spending function
Statistical Analysis 2: Comparison: Treme 300 mg x1 Dose + Durva 1500 mg vs Sora 400 mg; The analysis was performed using a Cox proportional hazards model adjusting for treatment, etiology of liver disease (HBV versus HCV versus others), ECOG (0 versus 1), and macro-vascular invasion (yes versus no). Values of the variables used for adjustment were obtained from IVRS; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.66 to 0.92]

2. Secondary Outcome: Overall Survival (OS) - Durva 1500 mg vs Sora 400 mg
Description: OS was defined as the time from the date of randomization until death due to any cause, regardless of whether the participant withdrew from randomized therapy or received another anticancer therapy. Any participant not known to have died at the DCO date was censored based on the last recorded date on which the participant was known to be alive. If the last known date alive or if the date of death was after the DCO date, participants were censored at the DCO date. This secondary outcome measure presents OS analysis of Durva 1500 mg vs Sora 400 mg at the time of the final analysis DCO (27Aug2021).
Time Frame: as for outcome 1
Population: The FAS included all participants who were randomized. T75+D arm was closed during study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 389 | 389 | 153 | 389
months | 16.56 [14.06 to 19.12] | 16.43 [14.16 to 19.58] | 16.36 [12.39 to 19.65] | 13.77 [12.25 to 16.13]
Statistical Analysis 1: Comparison: Durva 1500 mg vs Sora 400 mg; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-interiority for the comparison of arm Durva 1500 mg vs Sora 400 mg is declared if the upper limit of the two-sided alpha adjusted CI for HR is less than the NI margin of 1.08; Regression, Cox; Hazard Ratio (HR) = 0.86, 95.67% CI 2-sided [0.73 to 1.03] — The 95.67% confidence interval were derived based upon the exact number of OS events for each comparison using the Lan and DeMets approach that approximates the O'Brien Fleming spending function
Statistical Analysis 2: Comparison: Durva 1500 mg vs Sora 400 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Superiority was tested sequentially per protocol as non-inferiority was satisfied; p = 0.0674, Log Rank — The adjusted alpha levels (0.0433) for the two-sided superiority test were derived based upon the exact number of OS events for each comparison using the Lan and DeMets approach that approximates the O'Brien Fleming spending function

3. Secondary Outcome: Overall Survival (OS) at 18, 24, and 36 Months After Randomization
Description: Percentage of participants who were alive at fixed time points (18, 24, and 36 months) after randomization. The estimated percentage of survival along with the 95% confidence interval were calculated using Kaplan-Meier technique on the full analysis set.
Time Frame: At 18, 24, and 36 months post-randomization. Assessed at the final analysis DCO (27Aug2021).
Population: The FAS included all participants who were randomized. T75+D arm was closed during study.
Measure: Number (95% Confidence Interval); unit: percentage of survival
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 389 | 393 | 153 | 389
percentage of survival
  Survival rate at 18 months | 47.4 [42.4 to 52.3] | 48.7 [43.6 to 53.5] | 46.4 [38.4 to 54.1] | 41.5 [36.5 to 46.4]
  Survival rate at 24 months | 39.6 [34.8 to 44.5] | 40.5 [35.6 to 45.3] | 37.3 [29.6 to 44.9] | 32.6 [27.9 to 37.4]
  Survival rate at 36 months | 24.7 [20.0 to 29.8] | 30.7 [25.8 to 35.7] | 22.9 [16.6 to 29.8] | 20.2 [15.8 to 25.1]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS (per Response Evaluation Criteria in Solid Tumors, version 1.1 [RECIST 1.1] using Investigator assessments) was defined as the time from the date of randomization until the date of objective disease progression or death by any cause in the absence of progression, regardless of whether the patient withdrew from study treatment or received another anticancer therapy prior to progression. Progression (i.e., PD) was defined as a at least 20% increase in the sum of diameters of TLs, taking as reference the smallest previous sum of diameters (nadir) - this includes the baseline sum if that is the smallest on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm from nadir.
Time Frame: Tumor scans performed at baseline, every 8 weeks for the first 48 weeks following randomization, and every 12 weeks thereafter until RECIST 1.1-defined progression. Assessed up to DCO (27Aug2021, to a maximum of approximately 46 months)
Population: The FAS included all participants who were randomized. T75+D arm was closed during study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 389 | 393 | 153 | 389
months | 3.65 [3.19 to 3.75] | 3.78 [3.68 to 5.32] | 3.65 [2.79 to 4.86] | 4.07 [3.75 to 5.49]

5. Secondary Outcome: Time To Progression (TTP)
Description: TTP was defined as the time from randomization until objective tumor progression in the absence of death. If participants died without tumor progression, they were censored at the time of death.
Time Frame: From the date of randomization until objective tumor progression, assessed until the final analysis DCO (27Aug2021, to a maximum of approximately 46 months).
Population: The FAS included all participants who were randomized. T75+D arm was closed during study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 389 | 393 | 153 | 389
months | 3.75 [3.68 to 5.42] | 5.42 [3.81 to 5.62] | 3.75 [3.55 to 5.59] | 5.55 [5.13 to 5.75]

6. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR (per RECIST 1.1 as assessed by the Investigator) was defined as the number (%) of participants with at least 1 confirmed visit response of CR or PR until progression, or the last evaluable assessment in the absence of progression. Participants who go off treatment without progression, receive a subsequent therapy, and then respond will not be included as responders in the ORR. Complete response (ie., CR) was defined as disappearance of all target lesions (TLs) since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis diameter to <10 mm. Partial response (ie., PR) was defined as at least a 30% decrease in the sum of the diameter of TL, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 5
Population: The FAS included all participants who were randomized. T75+D arm was closed during study.
Measure: Count of Participants; unit: Participants
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 389 | 393 | 153 | 389
Participants | 66 | 79 | 26 | 20

7. Secondary Outcome: Disease Control Rate (DCR)
Description: Number (%) of participants with a Best Objective Response (BoR) of CR, PR, or SD. Complete response (ie., CR) was defined as disappearance of all target lesions (TLs) since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis diameter to <10 mm. Partial response (ie., PR) was defined as at least a 30% decrease in the sum of the diameter of TL, taking as reference the baseline sum of diameters. Stable disease (ie., SD) was defined as neither sufficient decrease in sum of diameters to qualify for PR nor sufficient increase to qualify for progression.
Time Frame: From the date of randomization until objective tumor progression or date of death, assessed until the final analysis DCO (27Aug2021, to a maximum of approximately 46 months).
Population: The FAS included all participants who were randomized. T75+D arm was closed during study.
Measure: Count of Participants; unit: Participants
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 389 | 393 | 153 | 389
Participants
  Yes | 213 | 236 | 89 | 236
  No | 176 | 157 | 64 | 153

8. Secondary Outcome: Duration of Objective Response (DoR)
Description: Time from the date of first documented confirmed response (complete or partial response) until the first date of documented progression or death in the absence of disease progression. Complete response (ie., CR) was defined as disappearance of all target lesions (TLs) since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis diameter to <10 mm. Partial response (ie., PR) was defined as at least a 30% decrease in the sum of the diameter of TL, taking as reference the baseline sum of diameters.
Time Frame: From the date of first documented response until the first date of documented progression or death, assessed until the final analysis DCO (27Aug2021, to a maximum of approximately 46 months).
Population: A subset of FAS subjects who achieve confirmed CR or PR as determined per RECIST 1.1 using Investigator assessment. T75+D arm was closed during study.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 66 | 79 | 26 | 20
months
  Duration of response from onset of response | 16.82 [7.43 to NA] — Not reached | 22.34 [8.54 to NA] — Not reached | 14.75 [7.46 to 14.75] | 18.43 [6.51 to 25.99]
  Time to onset of response from randomization | 2.09 [1.87 to 3.98] | 2.17 [1.84 to 3.98] | 2.02 [1.87 to 3.71] | 3.78 [1.89 to 8.44]

9. Secondary Outcome: Overall Survival (OS) by PD-L1
Description: Overall survival by baseline PD-L1 expression levels (positive vs. negative). PD-L1 expression level is based on the Tumor and Immune Cell Positivity (TIP) score method as: PD-L1 Positive (TIP ≥ 1%) or PD-L1 Negative (TIP < 1%).
Time Frame: From the date of randomization until death due to any cause, assessed until the final analysis DCO (27Aug2021, to a maximum of approximately 46 months).
Population: A subset of FAS who had non-missing baseline PD-L1 status. T75+D arm was closed during study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 344 | 337 | 144 | 329
months
  PD-L1 expression positive (TIP>=1%): number analyzed (Participants) | 154 | 148 | 65 | 148
  PD-L1 expression positive (TIP>=1%) | 17.22 [12.29 to 24.38] | 17.00 [13.11 to 22.31] | 24.21 [14.55 to 27.24] | 15.93 [10.68 to 21.72]
  PD-L1 expression negative (TIP<1%): number analyzed (Participants) | 190 | 189 | 79 | 181
  PD-L1 expression negative (TIP<1%) | 15.06 [12.68 to 18.53] | 14.26 [11.50 to 21.29] | 14.46 [8.97 to 17.51] | 13.93 [12.39 to 16.69]

10. Secondary Outcome: EORTC QLQ-C30 Time to Global Health Status/QoL Deterioration
Description: European Organisation for Research and Treatment of Cancer (EORTC) 30-item core quality of life questionnaire (QLQ-C30), which consists of 30 questions combined to produce a global health status/QoL scale. Higher scores indicate better health. A clinically meaningful deterioration is defined as a decrease in the score from baseline of ≥10. Time to deterioration is defined as the time from the date of randomization until the date of the first clinically meaningful deterioration that is confirmed at a subsequent visit or death by any cause in the absence of a clinically meaningful deterioration, regardless of whether the patient discontinues study drug(s) or receives another anticancer therapy.
Time Frame: At baseline and every 8 weeks for the first 48 weeks and then every 12 weeks thereafter until death or the final analysis DCO (27Aug2021), assessed up to approximately 46 months.
Population: A subset of the FAS who had baseline scores of >=10. T75+D arm was closed during study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 319 | 302 | 132 | 323
months | 7.4 [5.68 to 9.33] | 7.5 [5.82 to 10.84] | 7.3 [5.65 to 9.33] | 5.7 [4.80 to 7.39]

11. Secondary Outcome: EORTC QLQ-HCC18 Time to Symptom (Abdominal Pain) Deterioration
Description: EORTC 18-item hepatocellular cancer health-related quality of life questionnaire (QLQ-HCC18) is an 18-item questionnaire design used along with the 30-item EORTC QLQ-C30, which includes 8 symptom scales such as fatigue, jaundice, body image, nutrition, pain, fever, sex life and abdominal swelling. A high score for a symptom scale/item represents a high level of symptomatology/problem. A clinically meaningful deterioration is defined as an increase in the score from baseline of ≥10. Time to deterioration is defined as the time from the date of randomization until the date of the first clinically meaningful deterioration that is confirmed at a subsequent visit or death by any cause in the absence of a clinically meaningful deterioration, regardless of whether the patient discontinues study drug(s) or receives another anticancer therapy.
Time Frame: as for outcome 10
Population: A subset of the FAS who have a baseline symptom score <= 90. T75+D arm was closed during study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 315 | 291 | 127 | 314
months | 14.1 [9.46 to 24.41] | 16.8 [11.17 to NA] — Not reached | 14.7 [8.97 to 36.04] | 8.9 [7.23 to 11.14]

12. Secondary Outcome: EORTC QLQ-HCC18 Time to Symptom (Shoulder Pain) Deterioration
Description: as for outcome 11
Time Frame: as for outcome 10
Population: A subset of the FAS who have a baseline symptom score <= 90. T75+D arm was closed during study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 308 | 288 | 127 | 309
months | 16.0 [9.03 to 22.31] | 12.6 [9.23 to 19.58] | 13.8 [6.47 to 19.19] | 9.4 [7.46 to 13.37]

13. Secondary Outcome: EORTC QLQ-HCC18 Time to Symptom (Abdominal Swelling) Deterioration
Description: as for outcome 11
Time Frame: as for outcome 10
Population: A subset of the FAS who have a baseline symptom score <= 90. T75+D arm was closed during study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 314 | 290 | 125 | 319
months | 16.7 [9.46 to 24.8] | 20.9 [12.88 to 36.01] | 11.3 [5.78 to 19.19] | 11.1 [9.26 to 13.73]

14. Secondary Outcome: Presence of ADA for Durvalumab
Description: Number of participants with Anti-Drug Antibody (ADA) response to Durvalumab. ADA positive post-baseline only was also referred to as treatment-induced ADA. Treatment-emergent ADA was defined as the sum of treatment-induced ADA and treatment-boosted ADA. Results are reported as number of participants with ADA responses to Durvalumab for each indicated category.
Time Frame: Samples were collected on Day 1 (Week 0), Week 12 and at 3 months after the last dose of durvalumab. Assessed until the final analysis DCO (27Aug2021, to a maximum of approximately 46 months).
Population: The Durvalumab ADA evaluable set includes all participants who received at least 1 dose of Durvalumab and had non-missing baseline ADA and at least 1 non-missing post-baseline ADA results for Durvalumab. T75+D arm was closed during study.
Measure: Count of Participants; unit: Participants
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 282 | 294 | 108 | 0
Participants
  Treatment-emergent ADA positive (ADA Incidence) | 8 | 9 | 5 |
  Treatment-induced ADA (Positive Post-baseline only) | 7 | 9 | 5 |

15. Secondary Outcome: Presence of ADA for Tremelimumab
Description: Number of participants with Anti-Drug Antibody (ADA) response to Tremelimumab. ADA positive post-baseline only was also referred to as treatment-induced ADA. Treatment-emergent ADA was defined as the sum of treatment-induced ADA and treatment-boosted ADA. Results are reported as number of participants with ADA responses to Tremelimumab for each indicated category.
Time Frame: Samples were collected on Day 1 (Week 0), Week 12 and at 3 months after the last dose of tremelimumab. Assessed up to approximately 46 months after the first randomization.
Population: The Tremelimumab ADA evaluable set includes all participants who received at least 1 dose of Tremelimumab and had non-missing baseline ADA and at least 1 non-missing post-baseline ADA results for Tremelimumab. T75+D arm was closed during study.
Measure: Count of Participants; unit: Participants
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 0 | 182 | 102 | 0
Participants
  Treatment-emergent ADA positive (ADA Incidence) |  | 20 | 23 |
  Treatment-induced ADA (Positive Post-baseline only) |  | 20 | 22 |

16. Secondary Outcome: Summary of Durvalumab Concentration Over Time
Description: Blood sample were collected at pre-specified timepoints and Durvalumab concentrations in serum (ug/mL) were reported over time.
Time Frame: To evaluate the PK of Durvalumab, samples were collected pre-dose at week 4 and week 12 and post-dose at week 12. Assessed at the final analysis DCO (27Aug2021).
Population: PK analysis set includes all participants who received at least 1 dose Durvalumab per the study protocol for whom any PK post-dose data were available (ie, at least 1 non-missing post-dose PK result). T75+D arm was closed during study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 357 | 388 | 142 | 0
ug/mL
  Cycle 2 (Week 4) pre-dose, Geometric mean: number analyzed (Participants) | 340 | 314 | 142 | 0
  Cycle 2 (Week 4) pre-dose, Geometric mean | 74.7 (86.7) | 59.9 (101.6) | 65.1 (68.4) |
  Cycle 4 (Week 12) pre-dose, Geometric mean: number analyzed (Participants) | 252 | 253 | 142 | 0
  Cycle 4 (Week 12) pre-dose, Geometric mean | 113.9 (116.2) | 77.5 (280.1) | 92.1 (137.5) |
  Cycle 4 (Week 12) post-dose, Geometric mean: number analyzed (Participants) | 255 | 248 | 142 | 0
  Cycle 4 (Week 12) post-dose, Geometric mean | 556.9 (32.7) | 539.3 (38.6) | 528.4 (36.8) |

17. Secondary Outcome: Summary of Tremelimumab Concentration Over Time
Description: Blood sample were collected at pre-specified timepoints and Tremelimumab concentrations in serum (ug/mL) were reported over time.
Time Frame: To evaluate the PK of Tremelimumab, samples were collected at week 0 (post-dose), week 4, and week 12. Assessed at the final analysis DCO (27Aug2021).
Population: PK analysis set includes all participants who received at least 1 dose of Tremelimumab per the study protocol for whom any PK post-dose data were available (ie, at least 1 non-missing post-dose PK result). T75+D arm was closed during study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
Number analyzed (Participants) | 0 | 388 | 142 | 0
ug/mL
  Cycle 1 (Week 0) post-dose, Geometric mean: number analyzed (Participants) | 0 | 379 | 0 | 0
  Cycle 1 (Week 0) post-dose, Geometric mean |  | 78.0 (117.2) |  |
  Cycle 2 (Week 4), Geometric mean: number analyzed (Participants) | 0 | 221 | 132 | 0
  Cycle 2 (Week 4), Geometric mean |  | 10.7 (84.7) | 3.2 (67.8) |
  Cycle 4 (Week 12), Geometric mean: number analyzed (Participants) | 0 | 113 | 86 | 0
  Cycle 4 (Week 12), Geometric mean |  | 1.3 (156.5) | 4.3 (85.4) |

ADVERSE EVENTS:
Time Frame: All treatment-emergent adverse events (TEAEs) were collected up to the final analysis DCO (27Aug2021, to a maximum of approximately 46 months).
Description: TEAE was defined as any AE that started after dosing or prior to dosing and worsens following treatment exposure. AE was observed up until 90 days following discontinuation of the last dose of study drug, or until the initiation of the first subsequent therapy following discontinuation of treatment. All-cause mortality was reported for all randomized participants. Adverse events were reported for participants who received at least 1 dose of study drug regardless of the randomized assignment.
Arm/Group | Durva 1500 mg | Treme 300 mg x1 Dose + Durva 1500 mg | Treme 75 mg x4 Doses + Durva 1500 mg | Sora 400 mg
All-Cause Mortality (participants affected / at risk) | 280/389 | 262/393 | 123/153 | 293/389
Serious Adverse Events (participants affected / at risk) | 115/388 | 157/388 | 52/152 | 111/374
Other Adverse Events (participants affected / at risk) | 299/388 | 334/388 | 133/152 | 333/374
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durva 1500 mg (N=388) | Treme 300 mg x1 Dose + Durva 1500 mg (N=388) | Treme 75 mg x4 Doses + Durva 1500 mg (N=152) | Sora 400 mg (N=374)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatitis c (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis listeria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 7 (7) | 6 (6) | 8 (8)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 5 (5) | 3 (3) | 2 (2)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Glucocorticoid deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic wound (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 6 (6)
Bacillus bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune enteropathy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salmonella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 8 (8) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suspected covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post embolisation syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 4 (7) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 0 (0) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 (6) | 1 (2) | 3 (3) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 7 (9) | 0 (0) | 4 (5)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Internal haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 9 (9) | 4 (4) | 6 (6)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric varices haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 7 (8) | 0 (0) | 3 (4)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 8 (8) | 4 (4) | 5 (5) | 5 (5)
Dehiscence (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 4 (5) | 0 (0) | 2 (2)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 3 (3) | 3 (3) | 2 (2) | 5 (5)
Hepatic function abnormal (Hepatobiliary disorders) | 5 (6) | 1 (1) | 1 (1) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 3 (3) | 4 (4) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durva 1500 mg (N=388) | Treme 300 mg x1 Dose + Durva 1500 mg (N=388) | Treme 75 mg x4 Doses + Durva 1500 mg (N=152) | Sora 400 mg (N=374)
Alanine aminotransferase increased (Investigations) | 42 (49) | 35 (45) | 9 (9) | 20 (26)
Amylase increased (Investigations) | 9 (11) | 28 (38) | 6 (6) | 10 (17)
Aspartate aminotransferase increased (Investigations) | 54 (63) | 46 (53) | 16 (17) | 24 (33)
Blood bilirubin increased (Investigations) | 23 (30) | 19 (23) | 4 (5) | 29 (32)
Gamma-glutamyltransferase increased (Investigations) | 12 (12) | 18 (18) | 7 (7) | 19 (24)
Lipase increased (Investigations) | 23 (27) | 32 (38) | 8 (10) | 15 (17)
Decreased appetite (Metabolism and nutrition disorders) | 53 (58) | 65 (69) | 24 (24) | 67 (72)
Back pain (Musculoskeletal and connective tissue disorders) | 32 (35) | 28 (35) | 10 (11) | 13 (13)
Anaemia (Blood and lymphatic system disorders) | 28 (29) | 32 (39) | 13 (15) | 31 (32)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (11) | 10 (12) | 12 (14)
Insomnia (Psychiatric disorders) | 21 (21) | 40 (44) | 10 (10) | 16 (16)
Hyperthyroidism (Endocrine disorders) | 9 (9) | 30 (31) | 9 (10) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (34) | 30 (31) | 16 (19) | 22 (22)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 2 (2) | 26 (26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 23 (24) | 6 (6) | 14 (15)
Hypothyroidism (Endocrine disorders) | 19 (20) | 47 (47) | 19 (20) | 16 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 1 (1) | 53 (54)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 3 (3) | 173 (197)
Pruritus (Skin and subcutaneous tissue disorders) | 56 (61) | 89 (106) | 27 (34) | 24 (25)
Rash (Skin and subcutaneous tissue disorders) | 39 (51) | 84 (101) | 27 (32) | 50 (54)
Hypertension (Vascular disorders) | 17 (18) | 22 (26) | 6 (10) | 68 (79)
Abdominal pain upper (Gastrointestinal disorders) | 21 (24) | 29 (35) | 6 (9) | 18 (18)
Constipation (Gastrointestinal disorders) | 42 (48) | 36 (45) | 12 (13) | 34 (36)
Diarrhoea (Gastrointestinal disorders) | 57 (67) | 97 (125) | 28 (39) | 164 (241)
Dyspepsia (Gastrointestinal disorders) | 15 (17) | 9 (9) | 5 (5) | 20 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (18) | 15 (20) | 10 (14) | 22 (26)
Vomiting (Gastrointestinal disorders) | 18 (21) | 24 (28) | 8 (10) | 34 (37)
Asthenia (General disorders) | 48 (63) | 39 (46) | 20 (22) | 44 (49)
Fatigue (General disorders) | 37 (49) | 65 (71) | 25 (31) | 70 (75)
Oedema peripheral (General disorders) | 24 (25) | 32 (34) | 16 (18) | 19 (21)
Pyrexia (General disorders) | 31 (38) | 48 (62) | 16 (18) | 32 (34)
Weight decreased (Investigations) | 11 (12) | 28 (28) | 8 (8) | 36 (37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 (46) | 35 (38) | 11 (12) | 21 (21)
Abdominal pain (Gastrointestinal disorders) | 35 (36) | 44 (46) | 24 (26) | 59 (72)
Ascites (Gastrointestinal disorders) | 24 (26) | 22 (24) | 8 (8) | 20 (21)
Nausea (Gastrointestinal disorders) | 37 (41) | 46 (53) | 13 (13) | 52 (61)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 9 (11) | 0 (0) | 29 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees not to independently publish the results of the Study until first occurrence of one of the following: (i) multi-centre primary Publication is published; (ii) no multi-centre primary publication is submitted within two years after conclusion, abandonment, or termination of the Study at all sites; or (iii) Sponsor confirms in writing there will be no multi-centre primary Publication.

DOCUMENTS (2):
  • Study Protocol (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT03298451/Prot_016.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT03298451/SAP_018.pdf